CLINICAL TRIAL: NCT01325610
Title: The Effect of Oral Cholecalciferol (Vitamin D3) on Calcium Absorption in Persons on Long-term Hemodialysis
Brief Title: Vitamin D Effect on Calcium Absorption on Persons on Hemodialysis
Acronym: NEPH-Cal-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Principal Investigator, Laura Armas, Assistant Professor, Creighton University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #10-15975
Record Dates: First submitted 2011-01-17; First posted 2011-03-30 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease; Vitamin D Deficiency
Keywords: vitamin D; kidney; renal
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: cholecalciferol — a weekly dose of 20,000 IU of vitamin D3 will be given orally for 12 weeks.
  Other Names: Maximum D3, cholecalciferol, 10,000IU/capsule, 0.25mg USP, Pro-Pharma LLA, Kirksville, Mo

SUMMARY:
The assumption has been that 1,25(OH)2D is solely responsible for calcium absorption. That has been one of the presumed causes of hyperparathyroidism in chronic kidney disease (CKD) (low 1,25(OH)2D leads to decreased calcium absorption, which increases parathyroid hormone release in compensation). Replacing 1,25 D directly has been the goal with using 1,25D or its analogues in CKD. There is very little data concerning use of native vitamin D or 25(OH)D in CKD, although autocrine functions in extrarenal tissues would use 25(OH)D. The latest KDIGO guidelines do recognize the autocrine role of vitamin D, but have no data on outcomes or doses or optimal levels to guide them and so have made a blanket recommendation to treat 25D levels in CKD by general healthy population guidelines.

1. This project focuses on an outcome (calcium absorption) that may be impacted by optimizing 25D status in renal patients. The investigators will assume for this project that a level of 25D > 32 ng/ml is optimal in CKD patients as in a healthy population.
2. A secondary outcome is to quantify calcium absorption in CKD patients with and without vitamin D repletion and to quantify systemic 1,25D levels. This may clarify the roles 25D and 1,25D play in calcium absorption.

ELIGIBILITY:
Inclusion Criteria:

* on hemodialysis
* > 19 years of age

Exclusion Criteria:

* Pregnancy or planned pregnancy
* Hypercalcemia (> 10.2 mg/dl) at baseline
* Chronic GI disease
* Liver dysfunction
* Taking steroids
* Received any investigational drugs within 4 weeks
* Any allergy to vitamin D3
* Chronic vitamin D intake > 1,000 IU daily
* Dialysate concentration (calcium 2.5mg/L) which is to remain constant during Rx

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Vitamin D Status as measured by 25(OH)D levels | 12 weeks
  A weekly dose of 20,000 IU of vitamin D3 will be taken by the particpant and blood drawn to measure levels at weeks 1, 3, 5, 8, 10, 13, and 18.

SECONDARY OUTCOMES:
Calcium Absorption | 12 weeks
  A calcium absorption test will be done at baseline and after 12 weeks of vitamin D treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Laura AG Armas, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Graeff-Armas LA, Kaufmann M, Lyden E, Jones G. Serum 24,25-dihydroxyvitamin D3 response to native vitamin D2 and D3 Supplementation in patients with chronic kidney disease on hemodialysis. Clin Nutr. 2018 Jun;37(3):1041-1045. doi: 10.1016/j.clnu.2017.04.020. Epub 2017 Apr 30. PMID 28506446
- [Derived] Armas LA, Zena M, Lund R, Heaney RP. Calcium absorption response to cholecalciferol supplementation in hemodialysis. Clin J Am Soc Nephrol. 2013 Jun;8(6):1003-8. doi: 10.2215/CJN.08610812. Epub 2013 Feb 14. PMID 23411428